CLINICAL TRIAL: NCT07095322
Title: Women in Strength: A Randomised Pilot Feasibility Trial of a Muscle Strengthening Exercise Intervention for Women
Brief Title: Investigating the Feasibility and Acceptability of Co-created Intervention to Improve Women's Participation in Muscle-strengthening Exercises
Acronym: WISH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor Stuart Gray, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WISH
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Physical Activities; Exercise; Muscular Strength; Healthy Women
Keywords: Exercise; Muscle-strengthening; Women; Co-creation; co-design intervention; WISH study
MeSH Terms: conditions — Motor Activity | interventions — Educational Status; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Remain usual activity level
- Intervention (Experimental): Participated in the co-created intervention
  Interventions: Behavioral: Strength Education Session; Behavioral: Gym Membership; Behavioral: Group Exercise Session; Behavioral: Training Log; Behavioral: Support group

INTERVENTIONS:
Behavioral: Strength Education Session — Strength education session given at the first 4 weeks of intervention to educate women on muscle-strengthening exercises
  Other Names: Education
  Arms: Intervention
Behavioral: Gym Membership — 12 weeks gym membership to allow participant to go to the gym on their own
  Arms: Intervention
Behavioral: Group Exercise Session — Optional exercise sessions from week 4 to week 12 of the intervention if the participants want to join
  Other Names: Exercise session
  Arms: Intervention
Behavioral: Training Log — To record the exercise done for 24 weeks duration. Consist of date, day, exercise, set, repetitions, load, RPE
  Other Names: Log
  Arms: Intervention
Behavioral: Support group — For reminders and support for the participant for the first 12 weeks of intervention
  Arms: Intervention

SUMMARY:
This study will utilise the Randomised Controlled Trial (RCT) design. Following completion of the baseline measurements, participants will be randomly assigned to either the control group or the intervention group.

Control Group Control group will be asked to maintain normal activity levels for 24 weeks. On completion of the 24 weeks, 12-week University of Glasgow Sports gym membership will be given.

Intervention Group The overall aim of the intervention is for participants to participate in muscle strengthening exercises, of choice, two days a week. These exercises can include weight machine, resistance band and body weight resistance exercises, alongside strength training classes such as yoga and body pump. The intervention will begin with weekly education sessions over the first 4 weeks, to help make sure participants are confident and competent in performing exercises. Participants will be given a gym membership for the 12-week intervention period and asked to log all muscle strengthening exercises that participants participate in. Throughout the intervention, participants will receive weekly support reminder messages via WhatsApp from the research team, and researcher will also set up a social support group on WhatsApp for the participants. Weekly group-based exercise sessions with the researcher will also be offered to the participants; these will be optional.

The following data will be collected from all participants. All measures will be collected at baseline, mid-intervention measurement (week 6), post-intervention (week 12), and follow-up (week 24) except for follow-up interview and participants will be given an Amazon voucher worth £25 for every measurement period attend. Each test/measure is detailed further below.

During baseline measurement, researcher will ask the participants on their age, postcode, ethnic background, work situation, highest qualification completed, marital status, caregiver or not and the rating of health. Following this researcher will measure participants' body composition where the weight, height, fat mass, fat percentages, muscle mass and muscle size will be recorded.

Muscular strength will be measured using three strength tests which are the grip strength test, back strength test and maximal voluntary contraction. Participants will be shown how to perform the test by the research team before performing it. Participants will be asked to do each test 3 times with rest in between each attempt. The body composition and strength test will be conducted again in week 6, 12 and 24.

Intervention group will be involved in a follow-up interview during the measurement visit on week 12 and 24 to discuss the experiences and feedback on the intervention with the researchers.

ELIGIBILITY:
Inclusion Criteria:

* female
* between 18-45 years old
* living in Glasgow area
* not currently achieving the government recommendation of 2 days a week of muscle-strengthening activities

Exclusion Criteria:

* did not pass the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+)
* have blood pressure > 150/90 mmhg
* currently pregnant, planning to get pregnant within the next 6 months or in post-partum period in the past 6 months
* have intellectual disabilities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 31 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Interview with researcher on the feasibility and acceptability of the co-created intervention. | Week 12 (post intervention) - how they find the intervention Week 24 (follow up) - to see if they still continue participating in muscle-strengthening exercises, were there any challenges and what has helped them
  Participants is invited to an interview with the researcher to discuss their opinion of the intervention component and if it has helps them to start and continue participating in muscle-strengthening exercises. Interview conducted at two time point week 12 and week 24. Interview will be conducted either in-person or online through Microsoft Teams and will be audio recorded for analysis purpose.

SECONDARY OUTCOMES:
Knee Extensor Strength | changes from baseline to week 6, 12 and 24
  Knee extensor maximal torque during isometric MVC
Grip Strength | Changes from baseline to week 6, 12 and 24
  measured via handgrip dynamometer
Back Strength | Changes from baseline to week 6, 12 and 24
  measured via back strength dynamometer
Vastus lateralis muscle thickness | Changes from baseline to week 6, 12 and 24
  measured via ultrasound
Height | Recorded at baseline (Week 0)
  Height recorded using a stadiometer in centimetre at the beginning of the study.
Bodyweight | Changes from baseline to week 6, and 24.
  Changes in bodyweight, recorded in kilogram. Measured via body composition analyser
Body Mass Index (BMI) | Changes from baseline to week 6, 12, and 24
  Will be calculated from the bodyweight (in kilogram) and height (in meter) according to the BMI formula (kg/m^2).
Body Fat Mass | Changes from baseline to week 6, 12 and 24.
  Changes in body fat mass, recorded in kilogram. Measured via body composition analyser
Body Fat Percentages | Changes from baseline to week 6, 12, and 24
  Changes in body fat percentage, recorded in percentage. Measured via body composition analyser
Fat Free Mass | Changes from baseline to week 6, 12, and 24
  Changes in fat free mass, recorded in kilogram. Measured via body composition analyser

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No